CLINICAL TRIAL: NCT07170774
Title: Ischemic Preconditioning Enhances Aerobic Metabolic Energy Supply Capacity During Frequency Speed of Kick Test in Taekwondo Athletes: A Randomized Crossover Study
Brief Title: Research on the Enhancement of Aerobic Metabolic Energy Supply Capacity by Ischemic Preconditioning.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziyue Ou (Other)
Responsible Party: Sponsor-Investigator, Ziyue Ou, Sponsor-Investigator, Guangzhou Sport University
Organization: Guangzhou Sport University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2023WCXTD011
Record Dates: First submitted 2025-09-07; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Preconditioning; Aerobic Capacity
Keywords: Ischemic preconditioning; Energy metabolism; Sports performance; Oxygen uptake
MeSH Terms: interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPC Trial (Experimental): 220 mmHg
  Interventions: Device: Ischemic Preconditioning
- SHAM Trial (Placebo Comparator): 20 mmHg
  Interventions: Device: Sham

INTERVENTIONS:
Device: Ischemic Preconditioning — Compression cuff width: 10CM; Compression duration: 5min/5min (ischemia/reperfusion) *4. 220 mmHg
  Arms: IPC Trial
Device: Sham — Compression cuff width: 10CM; Compression duration: 5min/5min (compression/relaxation) *4. 20 mmHg
  Arms: SHAM Trial

SUMMARY:
The purpose of this clinical trial is to investigate whether IPC can improve aerobic capacity during exercise. The primary question it aims to answer is: Does IPC enhance the aerobic capacity of athletes? The researchers will compare IPC (220 mmHg pressure) with a placebo (20 mmHg pressure) to see if different interventions can enhance aerobic capacity and exercise performance.

Participants will:

* Undergo a randomized crossover controlled trial, visiting twice, with a one-week interval between each test.
* Conduct two assessments at the testing site each time, namely a pre-intervention assessment and a post-intervention assessment.
* Record their heart rate, blood pressure, weight, oxygen uptake, Taekwondo-specific performance, and other indicators.

ELIGIBILITY:
Inclusion Criteria:

* adult male athletes aged 18 years or older;
* taekwondo athletes classified as national second-class or above (having placed in the top three provincial professional taekwondo championships or the top eight national professional taekwondo championships);
* consistent and unified training over the past three months;
* no prior ischemic preconditioning;
* competitive taekwondo athletes.

Exclusion Criteria:

* supplementation with creatine;
* acute or chronic illnesses, including anxiety, depression, cardiovascular diseases, and metabolic disorders;
* engaging in vigorous physical activity within 48 hours prior to the experiment;
* consuming alcohol or caffeine within 24 hours before the experiment.

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Oxygen uptake | Participants had their oxygen uptake measured continuously during both visits, extending until six minutes after the completion of the exercise test.
  To record the oxygen uptake of the subjects and compare the changes in oxygen uptake after the intervention.
Taekwondo-specific sports performance test | The subjects rested quietly for five minutes before baseline measurements were taken. After this, the collection of metabolic gases commenced. Throughout the experiment, metabolic gases were continuously collected until six minutes after the tests.
  The specialized athletic ability in Taekwondo is measured by the number of kicks performed during the test.
Blood lactate | Blood lactate levels were measured at baseline, immediately after the intervention at 3 minutes, and at 3 and 10 minutes post-testing.
  Used to measure the intensity and metabolic adaptations during the testing process of taekwondo athletes

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Sport University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No
The data presented in this study are currently unpublished. The corresponding author will provide the relevant research data upon reasonable request after the associated paper has been officially accepted.

REFERENCES:
- [Background] Cheng CF, Kuo YH, Hsu WC, Chen C, Pan CH. Local and Remote Ischemic Preconditioning Improves Sprint Interval Exercise Performance in Team Sport Athletes. Int J Environ Res Public Health. 2021 Oct 12;18(20):10653. doi: 10.3390/ijerph182010653. PMID 34682399
- [Background] Chen Y, Yang J, Muradov O, Li X, Lee JKW, Qiu J. Effect of ischemic preconditioning on maximum accumulated oxygen deficit in 400-meter runners. Eur J Sport Sci. 2023 May;23(5):789-796. doi: 10.1080/17461391.2022.2064769. Epub 2022 Apr 25. PMID 35400298
- [Background] Caru M, Levesque A, Lalonde F, Curnier D. An overview of ischemic preconditioning in exercise performance: A systematic review. J Sport Health Sci. 2019 Jul;8(4):355-369. doi: 10.1016/j.jshs.2019.01.008. Epub 2019 Jan 23. PMID 31333890
- [Background] Albuquerque MR, Flor CAG, Ribeiro AIS, Mesquita PHC, Franchini E, Laurentino GC. Effects of Ischemic Preconditioning on Sport-Specific Performance in Highly Trained Taekwondo Athletes. Sports (Basel). 2024 Jun 26;12(7):179. doi: 10.3390/sports12070179. PMID 39058070